CLINICAL TRIAL: NCT05199675
Title: Implementing Digital Peer Support Training for Adolescent Mental Health: Study Protocol For A Type III Hybrid Randomized Controlled Trial
Brief Title: Implementing Digital Peer Support Training for Adolescent Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The N.1 Institute for Health (N.1) (Other)
Collaborators: Manjusri Secondary School, Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NUS-IRB-2021-761
Record Dates: First submitted 2021-12-15; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Adolescent Development; Peer Group; Mental Health Wellness 1
Keywords: Hybrid III trial,; Adolescence; Digital peer support; Mental Health; Implementation Science; Communication Science; Developmental psychology
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Using a hybrid type III trial with a cluster randomized design, a total of 100 Singaporean students from 4 classes in a high school will be randomly allocated to the intervention or wait-list control arm. The intervention arm will undergo bite size modules on the four active ingredients of youth mental well-being-specifically, Mattering, selfhood, compassion and mindfulness, which will be delivered through training workshops, simulation activities, and homework assignments. Students in the wait-list control arm will receive the the training program after the conclusion of the trial with the intervention arm. The pre-post with control evaluation design will be utilized to evaluate program outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Peer Support Training Program (Experimental): The intervention arm will undergo bite size modules on the four active ingredients of youth mental well-being-specifically, Mattering, selfhood, compassion and mindfulness, which will be delivered through training workshops, simulation activities, and homework assignments. The pre-post with control evaluation design will be utilized to evaluate program outcomes. Fidelity will be the primary outcome assessed to demonstrate the effectiveness of the digital peer support training program. It will be measured by the extent to which adolescents' responses to real-cases of peer disclosure indicate Mattering, selfhood, compassion and mindfulness. Reach, acceptability, cost-effectiveness, and adolescent self-reported psychological well-being will be assessed as secondary outcomes. Cost-effectiveness analysis will inform the development of a scalability and sustainability plan.
  Interventions: Behavioral: Digital Peer Support Training Program
- Waitlist control for Digital Peer Support Training Program (Active Comparator): Students in the wait-list control arm will receive the training program after the conclusion of the trial with the intervention arm. The pre-post with control evaluation design will be utilized to evaluate program outcomes. The intervention arm will undergo bite size modules on the four active ingredients of youth mental well-being-specifically, Mattering, selfhood, compassion and mindfulness, which will be delivered through training workshops, simulation activities, and homework assignments.The same set of primary and secondary outcomes assessed in the experimenter arm will be included. Specifically, fidelity will be the primary outcome assessed. Reach, acceptability, cost-effectiveness, and adolescent self-reported psychological well-being will be assessed as secondary outcomes.
  Interventions: Behavioral: Digital Peer Support Training Program

INTERVENTIONS:
Behavioral: Digital Peer Support Training Program — The digital peer support training program will consist of bite size modules on the four active ingredients of youth mental well-being, which will be delivered through training workshops, simulation activities, and homework assignments. The training will be conducted over 8 sessions, each lasting for 45-60 minutes following the typical duration of a school lesson on Character and Citizenship Education. The training workshops will be conducted as part of the school's Character and Citizenship Education lessons. The proficiency of participants in applying these digital support skills will be evaluated through simulation and homework activities, in which they apply the four active ingredients in their responses to mock letters that are adapted from actual cases of peer emotional disclosure. At the end of the training, adolescents are expected to apply the four active ingredients to the homework assignments on peers' emotional experiences.

SUMMARY:
Using a hybrid type III trial with a cluster randomized design, the digital peer support training for adolescent mental health protocol aims to implement a multidisciplinary program, which translates theoretical and empirical work from implementation science, communication science, and developmental psychology, to train adolescents in effective digital peer support for mental well-being.

With the lack of theoretically driven and empirically grounded program to train adolescents in providing digital peer support for mental well-being, this study involves the design and implementation of such a program using that addressed four research questions:

(a) what is digital peer support for adolescents, (b) how do peers provide effective peer support online, (c) how do we implement digital peer support training among adolescents, (d) what are the facilitators and barriers in training adolescents to provide effective peer support, and (e) how do we scale up and sustain digital peer support training among adolescents for far-reaching and long-lasting effectiveness?

DETAILED DESCRIPTION:
Background: The digital peer support training for adolescent mental health project aims to implement a multidisciplinary program, which translates theoretical and empirical work from implementation science, communication science, and developmental psychology, to train adolescents in effective digital peer support for mental well-being. Nearly 50% of all mental health issues has an early onset in adolescence, and mental health conditions have long lasting and far-reaching effects for adolescents. Although there is an emerging body of work that underscores digital platform as an important interpersonal context for peer support in managing well-being in adolescence, there is no implementation of an evidence-based intervention to train adolescents in effective online peer support.

Methods: Using a hybrid type III trial with a cluster randomized design, a total of 100 Singaporean students from 4 classes in a high school will be randomly allocated to the intervention or wait-list control arm. The intervention arm will undergo bite size modules on the four active ingredients of youth mental well-being-specifically, Mattering, selfhood, compassion and mindfulness, which will be delivered through training workshops, simulation activities, and homework assignments. Students in the wait-list control arm will receive the the training program after the conclusion of the trial with the intervention arm. The pre-post with control evaluation design will be utilized to evaluate program outcomes. Fidelity will be the primary outcome assessed to demonstrate the effectiveness of the digital peer support training program. It will be measured by the extent to which adolescents' responses to real-cases of peer disclosure indicate Mattering, selfhood, compassion and mindfulness. Reach, acceptability, cost-effectiveness, and adolescent self-reported psychological well-being will be assessed as secondary outcomes. Cost-effectiveness analysis will inform the development of a scalability and sustainability plan.

Data Collection, Management and Analyses: We conducted power analysis using to ascertain the adequate sample size needed for the randomized controlled trial, specifically in comparing the intervention and control groups on different implementation and clinical outcomes, so that the study has sufficient power to detect valid effects. The study sample size of n = 50 for intervention and n = 50 for control is needed because of multiple dependent variables measuring implementation outcomes included in the study--specifically, fidelity, reach, acceptability, and cost-effectiveness, and the testing of the clinical outcome on psychological well-being.

Missing data In dealing with missing data, we will determine if missing data is missing completely at random. If missing data is not systematic, as indicated by the non-significant result from Little's Missing Completely at Random Test, we will handle missing data using full information maximum likelihood imputation.

Qualitative analysis We will conduct qualitative analyses with NVivo 10 on the secondary outcome on acceptability of the program. This outcome data will be gathered from both the adolescents and their teachers using focus group discussions post-intervention to elucidate the facilitators and barriers at the individual and organization levels that contribute to and hinder adolescents in providing effective digital peer support, respectively. Participants' responses will be subjected to topic modelling using Latent Dirichlet Allocation (LDA) analyses with R to filter the huge amount of data available and drill down relevant themes and topics. LDA is an advanced statistical method that increases precision and accuracy in coding.

Quantitative analysis The paired-sample t test for continuous variables will be conducted with the intervention group to compare the pre- (i.e., first time point) and post-training scores (second time point) for the four active ingredients and we expect that the change score will be significant. Likewise, for the wait-list control group, their scores for the same two time-points will be assessed and it is expected that the change score will not be significant. The independent sample t-tests will be conducted to compare the intervention and control groups' scores at the first and second time points. For the first time point, we anticipate the difference between the intervention and control groups to be non-significant. Participants in both arms are expected to have comparable initial level of digital peer support skills-specifically, their knowledge of and competency in harnessing the four active ingredients in responding to real cases of peer disclosure. On the contrary, for the second time point, the difference between the intervention and control groups is anticipated to be significant, with the former indicating a higher composite score of effective peer support, if the digital peer support training program is effective.

Discussion: The digital peer support training trial adopts a multidisciplinary approach to implement a theoretically grounded and evidence-based practice for training adolescents to be effective peer supporters online-an important precursor in implementing relevant and impactful digital peer support intervention for youth mental well-being.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include certified teachers aged 22 to 65 with a post-graduate diploma in education and who teach the Character and Citizenship Education lessons, as well as adolescents aged 13 to 16 who are students enrolled in the high school.

Exclusion Criteria:

* Students who have been identified by the school teachers and counselors prior to the training as experiencing emotional distress will be excluded. Additionally, as one of the secondary outcomes examined in this study, students with low ratings of psychological well-being (Ryff & Keyes, 1995; i.e., 2 SD below the mean) in the pre-training assessment will be referred to the teachers and school counselors and they will not participate in the workshop.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fidelity--Mattering | Before and immediately after training (as pre-class activity and homework assignment, respectively)
  The degree to which the program is delivered as intended--specifically, fidelity will be measured by the extent to which adolescents' responses to real-world cases of peer disclosure indicate Mattering, using the 5-item Rosenberg Mattering Scale (Rosenberg & McCullough, 1981) on a 5-point scale 0 (not at all) to 4 (very much).
  Before and immediately after training (as pre-class activity and homework assignment, respectively), participants in both the intervention arm will be presented with three cases of peer disclosure of varying levels of complexity and social context/issues (i.e., family, school, and relationship).
Change in Fidelity--Selfhood | Before and immediately after training (as pre-class activity and homework assignment, respectively)
  The degree to which the program is delivered as intended--specifically, fidelity will be measured by the extent to which adolescents' responses to real-world cases of peer disclosure indicate selfhood using the 10-item Rosenberg Global Self-Esteem Scale (Rosenberg, 1989), rated on a 5-point scale 0 (not at all) to 4 (very much).
  Before and immediately after training (as pre-class activity and homework assignment, respectively), participants in both the intervention arm will be presented with three cases of peer disclosure of varying levels of complexity and social context/issues (i.e., family, school, and relationship).
Change in Fidelity--compassion | Before and immediately after training (as pre-class activity and homework assignment, respectively)
  The degree to which the program is delivered as intended--specifically, fidelity will be measured by the extent to which adolescents' responses to real-world cases of peer disclosure indicate compassion as operationalized in the Compassion Cultivation Training protocol (Jazaieri et al., 2013) as a multidimensional process comprising of four key components. Each component will be rated on a 5-point scale 0 (not at all) to 4 (very much).
  Before and immediately after training (as pre-class activity and homework assignment, respectively), participants in both the intervention arm will be presented with three cases of peer disclosure of varying levels of complexity and social context/issues (i.e., family, school, and relationship).
Change in Fidelity--Mindfulness | Before and immediately after training (as pre-class activity and homework assignment, respectively)
  The degree to which the program is delivered as intended--specifically, fidelity will be measured by the extent to which adolescents' responses to real-world cases of peer disclosure indicate indicate mindfulness using the Cognitive theory of mindfulness(Carson & Langer, 2006). Participants' responses will be evaluated based on the extent in which they reflect/harness the techniques for enhancing mindful self-acceptance in their responses using a 5-point scale 0 (not at all) to 4 (very much).
  Before and immediately after training (as pre-class activity and homework assignment, respectively), participants in both the intervention arm will be presented with three cases of peer disclosure of varying levels of complexity and social context/issues (i.e., family, school, and relationship).

SECONDARY OUTCOMES:
Reach | Immediately after the training program/last session of the training workshop
  The number of adolescents who received the training divided by the number of eligible adolescents from the four classes (clusters), will be established.
Acceptability--Self-report | Immediately after the training program/last session of the training workshop
  We will measure acceptability from the perspective of both adolescents and their teachers using a self-report questionnaire post-intervention-specifically, at the last session of the training program.
  Participants will provide responses to the Client Satisfaction Questionnaire (CSQ-8; Attkisson & Greenfield, 1994), with 8 items that measure the degree of client satisfaction with services and will be rated on a 4-point scale ranging from 1 (poor) to 4 (excellent).
Acceptability--focus group discussions | Immediately after the training program/last session of the training workshop
  We will measure acceptability from the perspective of both adolescents and their teachers using focus group discussions post-intervention-specifically at the last session of the training program, which will be audio-recorded and transcribed using pseudonyms to ensure confidentiality.
  Following the implementation steps delineated in the GTO framework (Wandersman et al., 2000), the focus group interviews with groups of 3 to 4 participants will elucidate facilitators and barriers at the individual level-specifically, factors that contribute to or hinder adolescents in providing effective digital peer support. At the organizational level, we will assess the fit of the training program within the school context by addressing the four primary questions listed earlier in the section on program implementation
Cost-effectiveness | Immediately after the training program/last session of the training workshop
  To estimate the cost of implementing the training program, which functions as important information for the research team as well as the participating organization in assessing the resources needed to scale up and sustain the program within the school system. The cost analysis will include different component of the implementation strategy, such as designing and improving the training program, conducting the training and the associated activities, participating adolescents' self-reported psychological well-being pre- and post-intervention, and their continued efficacy in providing digital peer support three and six months post-intervention.
Psychological well-being | Immediately after the training program/last session of the training workshop
  Adolescents' psychological well-being will be assessed using the 18-item Ryff's psychological well-being measure (Ryff & Keyes, 1995) on a 6-point scale that ranges from 1 (strongly disagree) to 6 (strongly agree). The measure consists of six dimensions, including positive relations with others, autonomy, environment mastery, personal growth, purpose in life, and self-acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: GeckHong Yeo, PhD, Principal Investigator — N.1 Institute for Health, National University of Singapore; Dean Ho, PhD, Principal Investigator — N.1 Institute for Health, National University of Singapore; Wei Ning Chang, PhD, Principal Investigator — Institute of Mental Health, Singapore; Bradford Brown, PhD, Principal Investigator — University of Wiscosnsin, Madison; Department of Educational Psychology

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in article publication, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 12 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose-for individual participant data meta-analysis. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Background] Kieling C, Baker-Henningham H, Belfer M, Conti G, Ertem I, Omigbodun O, Rohde LA, Srinath S, Ulkuer N, Rahman A. Child and adolescent mental health worldwide: evidence for action. Lancet. 2011 Oct 22;378(9801):1515-25. doi: 10.1016/S0140-6736(11)60827-1. Epub 2011 Oct 16. PMID 22008427
- [Background] Larson RW, Moneta G, Richards MH, Wilson S. Continuity, stability, and change in daily emotional experience across adolescence. Child Dev. 2002 Jul-Aug;73(4):1151-65. doi: 10.1111/1467-8624.00464. PMID 12146740
- [Background] Marques de Miranda D, da Silva Athanasio B, Sena Oliveira AC, Simoes-E-Silva AC. How is COVID-19 pandemic impacting mental health of children and adolescents? Int J Disaster Risk Reduct. 2020 Dec;51:101845. doi: 10.1016/j.ijdrr.2020.101845. Epub 2020 Sep 10. PMID 32929399
- [Background] Nearchou F, Flinn C, Niland R, Subramaniam SS, Hennessy E. Exploring the Impact of COVID-19 on Mental Health Outcomes in Children and Adolescents: A Systematic Review. Int J Environ Res Public Health. 2020 Nov 16;17(22):8479. doi: 10.3390/ijerph17228479. PMID 33207689
- [Background] Prinstein, M. J., & Giletta, M. (2016). Peer relations and developmental psychopathology. In D. Cicchetti (Ed.), developmental psychopathology (pp. 1-53). Hoboken, NJ: Wiley. https ://doi.org/10.1002/97811 19125 556.devps y112.
- [Background] Choukas-Bradley, S., & Prinstein, M. J. (2014). Peer relationships and the development of psychopathology. In M. Lewis & K. D. Rudolph (Eds.), Handbook of developmental psychopathology (pp. 185-204). Boston, MA: Springer
- [Background] Parker, J. (2006). Peer relationships, child development, and adjustment: A developmental psychopathology perspective. Developmental Psychopathology, Theory and Method, 1, 419. https://doi.org/10.1002/97804 70939 383.ch12.
- [Background] Valkenburg, P. M., & Peter, J. (2009). The effects of instant messaging on the quality of adolescents' existing friendships: A longitudinal study. Journal of Communication, 59, 79-97. http://dx.doi.org/10.1111/j.1460-2466.2008.01405.x
- [Background] Valkenburg PM, Peter J. Online communication among adolescents: an integrated model of its attraction, opportunities, and risks. J Adolesc Health. 2011 Feb;48(2):121-7. doi: 10.1016/j.jadohealth.2010.08.020. Epub 2010 Dec 13. PMID 21257109
- [Background] Choi, M., & Toma, C. L. (2014). Social sharing through interpersonal media: Patterns and effects on emotional well-being. Computers in Human Behavior, 36, 530-541. http://dx.doi.org/10.1016/j.chb.2014.04.026
- [Background] Huckins JF, daSilva AW, Wang W, Hedlund E, Rogers C, Nepal SK, Wu J, Obuchi M, Murphy EI, Meyer ML, Wagner DD, Holtzheimer PE, Campbell AT. Mental Health and Behavior of College Students During the Early Phases of the COVID-19 Pandemic: Longitudinal Smartphone and Ecological Momentary Assessment Study. J Med Internet Res. 2020 Jun 17;22(6):e20185. doi: 10.2196/20185. PMID 32519963
- [Background] Loades ME, Chatburn E, Higson-Sweeney N, Reynolds S, Shafran R, Brigden A, Linney C, McManus MN, Borwick C, Crawley E. Rapid Systematic Review: The Impact of Social Isolation and Loneliness on the Mental Health of Children and Adolescents in the Context of COVID-19. J Am Acad Child Adolesc Psychiatry. 2020 Nov;59(11):1218-1239.e3. doi: 10.1016/j.jaac.2020.05.009. Epub 2020 Jun 3. PMID 32504808
- [Background] Lippke S, Fischer MA, Ratz T. Physical Activity, Loneliness, and Meaning of Friendship in Young Individuals - A Mixed-Methods Investigation Prior to and During the COVID-19 Pandemic With Three Cross-Sectional Studies. Front Psychol. 2021 Feb 2;12:617267. doi: 10.3389/fpsyg.2021.617267. eCollection 2021. PMID 33603702
- [Background] Nesi J, Choukas-Bradley S, Prinstein MJ. Transformation of Adolescent Peer Relations in the Social Media Context: Part 1-A Theoretical Framework and Application to Dyadic Peer Relationships. Clin Child Fam Psychol Rev. 2018 Sep;21(3):267-294. doi: 10.1007/s10567-018-0261-x. PMID 29627907
- [Background] Fortuna KL, Venegas M, Umucu E, Mois G, Walker R, Brooks JM. The Future of Peer Support in Digital Psychiatry: Promise, Progress, and Opportunities. Curr Treat Options Psychiatry. 2019 Sep;6(3):221-231. doi: 10.1007/s40501-019-00179-7. Epub 2019 Jun 20. PMID 33796435
- [Background] Tolley JA, Michel MA, Williams AE, Renschler JS. Peer Support in the Treatment of Chronic Pain in Adolescents: A Review of the Literature and Available Resources. Children (Basel). 2020 Sep 7;7(9):129. doi: 10.3390/children7090129. PMID 32906581
- [Background] Gillard S. Peer support in mental health services: where is the research taking us, and do we want to go there? J Ment Health. 2019 Aug;28(4):341-344. doi: 10.1080/09638237.2019.1608935. Epub 2019 May 9. No abstract available. PMID 31070066
- [Background] Ramchand R, Ahluwalia SC, Xenakis L, Apaydin E, Raaen L, Grimm G. A systematic review of peer-supported interventions for health promotion and disease prevention. Prev Med. 2017 Aug;101:156-170. doi: 10.1016/j.ypmed.2017.06.008. Epub 2017 Jun 8. PMID 28601621
- [Background] Hart LM, Morgan AJ, Rossetto A, Kelly CM, Mackinnon A, Jorm AF. Helping adolescents to better support their peers with a mental health problem: A cluster-randomised crossover trial of teen Mental Health First Aid. Aust N Z J Psychiatry. 2018 Jul;52(7):638-651. doi: 10.1177/0004867417753552. Epub 2018 Feb 8. PMID 29417834
- [Background] Ali K, Farrer L, Gulliver A, Griffiths KM. Online Peer-to-Peer Support for Young People With Mental Health Problems: A Systematic Review. JMIR Ment Health. 2015 May 19;2(2):e19. doi: 10.2196/mental.4418. eCollection 2015 Apr-Jun. PMID 26543923
- [Background] Finding the next generation of mental health treatments and approaches. Wellcome.org. URL: https://wellcome.org/news/finding-next-generation-mental-health-treatments-and-approaches [access 2021-11-01]
- [Background] Marshall SK. Do I matter? Construct validation of adolescents' perceived mattering to parents and friends. J Adolesc. 2001 Aug;24(4):473-90. doi: 10.1006/jado.2001.0384. PMID 11549327
- [Background] Marshall SK. Relative contributions of perceived mattering to parents and friends in predicting adolescents' psychological well-being. Percept Mot Skills. 2004 Oct;99(2):591-601. doi: 10.2466/pms.99.2.591-601. PMID 15560349
- [Background] Marshall SK, Tilton-Weaver L. Adolescents' perceived mattering to parents and friends: testing cross-lagged associations with psychosocial well-being. International Journal of Behavioral Development 2019 Nov; 43(6):541-52. [doi: 10.1177/0165025419844019]
- [Background] Elliott G, Kao S, Grant AM. Mattering: empirical validation of a social-psychological concept. Self and Identity 2004 Oct 1; 3(4):339-54. [doi: 10.1080/13576500444000119]
- [Background] Baumeister RF. The self. In Finkel EJ, Baumeister RF, editors. Advanced social psychology: the state of the science. New York: Oxford University Press; 2016. p. 89-116. ISBN: 9780195381207
- [Background] Butzer, B., & Kuiper, N. A. (2006). Relationships between the frequency of social comparisons and self-concept clarity, intolerance of uncertainty, anxiety, and depression. Personality and Individual Differences 41(1), 167-176. https ://doi.org/10.1016/j.paid.2005.12.017.
- [Background] Flett GL, Nepon T. Mattering versus self-esteem in university students: associations with regulatory focus, social feedback, and psychological distress. Journal of Psychoeducational Assessment 2020 Sep; 38(6):663-74. [doi: 10.1177/0734282919890786]
- [Background] Van Gordon W, Shonin E, Griffiths MD. Towards a second generation of mindfulness-based interventions. Aust N Z J Psychiatry. 2015 Jul;49(7):591-2. doi: 10.1177/0004867415577437. Epub 2015 Mar 23. No abstract available. PMID 25801660
- [Background] Kirby JN, Tellegen CL, Steindl SR. A Meta-Analysis of Compassion-Based Interventions: Current State of Knowledge and Future Directions. Behav Ther. 2017 Nov;48(6):778-792. doi: 10.1016/j.beth.2017.06.003. Epub 2017 Jun 21. PMID 29029675
- [Background] Oberle E, Schonert-Reichl KA, Thomson KC. Understanding the link between social and emotional well-being and peer relations in early adolescence: gender-specific predictors of peer acceptance. J Youth Adolesc. 2010 Nov;39(11):1330-42. doi: 10.1007/s10964-009-9486-9. Epub 2009 Nov 29. PMID 20091211
- [Background] Nixon CL. Current perspectives: the impact of cyberbullying on adolescent health. Adolesc Health Med Ther. 2014 Aug 1;5:143-58. doi: 10.2147/AHMT.S36456. eCollection 2014. PMID 25177157
- [Background] Pavarini G, Reardon T, Hollowell A, Bennett V, Lawrance E; Peer Support Young People's Advisory Group; Pinfold V, Singh I. Online peer support training to promote adolescents' emotional support skills, mental health and agency during COVID-19: Randomised controlled trial and qualitative evaluation. Eur Child Adolesc Psychiatry. 2023 Jun;32(6):1119-1130. doi: 10.1007/s00787-021-01933-0. Epub 2022 Feb 17. PMID 35174419
- [Background] Wandersman, A., Imm, P., Chinman, M., & Kaftarian, S. (2000). Getting to outcomes: A results-based approach to accountability. Evaluation and program planning, 23(3), 389-395. https://doi.org/10.1016/S0149-7189(00)00028-8
- [Background] Albers, B., Mildon, R., Lyon, A. R., & Shlonsky, A. (2017). Implementation frameworks in child, youth and family services-Results from a scoping review. Children and Youth Services Review, 81, 101-116. https://doi.org/10.1016/j.childyouth.2017.07.003
- [Background] Ryff CD, Keyes CL. The structure of psychological well-being revisited. J Pers Soc Psychol. 1995 Oct;69(4):719-27. doi: 10.1037//0022-3514.69.4.719. PMID 7473027
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Miyamoto Y, Uchida Y, Ellsworth PC. Culture and mixed emotions: co-occurrence of positive and negative emotions in Japan and the United States. Emotion. 2010 Jun;10(3):404-15. doi: 10.1037/a0018430. PMID 20515228
- [Background] Ma X, Tamir M, Miyamoto Y. A socio-cultural instrumental approach to emotion regulation: Culture and the regulation of positive emotions. Emotion. 2018 Feb;18(1):138-152. doi: 10.1037/emo0000315. Epub 2017 Apr 17. PMID 28414476
- [Background] Rosenberg, M., & McCullough, B. C. (1981). Mattering: Inferred significance and mental health among adolescents. Research in Community & Mental Health, 2, 163-182.
- [Background] Rosenberg, M. (1989). Society and the adolescent self-image. Middleton, CT: Wesleyan University Press.
- [Background] Carson SH, Langer EJ. Mindfulness and self-acceptance. Journal of rational-emotive and cognitive-behavior therapy. 2006; 24(1):29-43.
- [Background] Attkisson, C. C., & Greenfield, T. K. (1994). Client Satisfaction Questionnaire-8 and Service Satisfaction Scale-30. In M. E. Maruish (Ed.), The use of psychological testing for treatment planning and outcome assessment (pp. 402-420). Lawrence Erlbaum Associates, Inc.
- [Background] Albers B, Shlonsky A, Mildon R, editors. Implementation Science 3.0. Springer Nature; 2020 Mar 18.
- [Background] QSR International. (2012). NVivo 10 [Computer software]. Retrieved from http://www.qsrinternational.com
- [Background] Richardson, G. M., Bowers, J., Woodill, A. J., Barr, J. R., Gawron, J. M., & Levine, R. A. (2014). Topic models: A tutorial with R. International Journal of Semantic Computing, 8, 85-98. https://doi.org/10.1142/S1793351X14500044
- [Background] Odgers CL, Jensen MR. Annual Research Review: Adolescent mental health in the digital age: facts, fears, and future directions. J Child Psychol Psychiatry. 2020 Mar;61(3):336-348. doi: 10.1111/jcpp.13190. Epub 2020 Jan 17. PMID 31951670
- [Background] Moir F, Henning M, Hassed C, Moyes SA, Elley CR. A Peer-Support and Mindfulness Program to Improve the Mental Health of Medical Students. Teach Learn Med. 2016 Jul-Sep;28(3):293-302. doi: 10.1080/10401334.2016.1153475. Epub 2016 Apr 19. PMID 27092397
- [Background] Huang J, Nigatu YT, Smail-Crevier R, Zhang X, Wang J. Interventions for common mental health problems among university and college students: A systematic review and meta-analysis of randomized controlled trials. J Psychiatr Res. 2018 Dec;107:1-10. doi: 10.1016/j.jpsychires.2018.09.018. Epub 2018 Sep 29. PMID 30300732
- [Background] Jazaieri H, Jinpa GT, McGonigal K, Rosenberg EL, Finkelstein J, Simon-Thomas E, Cullen M, Doty JR, Gross JJ, Goldin PR. Enhancing compassion: A randomized controlled trial of a compassion cultivation training program. Journal of Happiness Studies. 2013 Aug;14(4):1113-26. https://doi.org/10.1007/s10902-012-9373-z